CLINICAL TRIAL: NCT00783445
Title: Community Exercise and Metabolic Syndrome in Black Families
Brief Title: Evaluating the Effectiveness of a Community Exercise Program to Reduce the Risk of Metabolic Syndrome Among Black Americans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr. Diane Becker, Professor, Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 610; R01HL089474-01 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Cardiovascular Syndrome; Metabolic Syndrome; Obesity; Hyperglycemia
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Exercise in a community setting while supervised by a coach
  Interventions: Behavioral: Community-Based Exercise Program (C-FIT)
- 2 (Active Comparator): Self-exercise plan based on an individualized prescription after an initial fitness evaluation
  Interventions: Behavioral: Self-Help Exercise Program (HOME)

INTERVENTIONS:
Behavioral: Community-Based Exercise Program (C-FIT) — Participants will do 1 hour of exercise two to three times each week in a community setting for 1 year, while being supervised by a personal coach.
  Arms: 1
Behavioral: Self-Help Exercise Program (HOME) — After a fitness evaluation, participants will be given an exercise prescription and recommendations for home-based, self-mediated progressive exercise. Participants will be expected to do 1 hour of exercise two to three times each week for 1 year.
  Arms: 2

SUMMARY:
Black Americans with a family history of early heart disease tend to have a group of risk factors that can contribute to heart disease. These risk factors, which include excess body weight, high blood pressure, and high cholesterol, are known collectively as metabolic syndrome. This study will compare a community-based, coach-led exercise program to an individual, self-led home-based exercise program to determine which program is more effective at reducing the metabolic syndrome risk factors that can lead to heart disease.

DETAILED DESCRIPTION:
Metabolic syndrome is a term that is used to describe a group of risk factors for coronary artery disease (CAD). The risk factors include abdominal obesity, insulin resistance, high cholesterol, and high blood pressure. People who live a sedentary lifestyle and do not get enough exercise are at risk of developing metabolic syndrome and CAD. Black Americans also have an increased risk of metabolic syndrome and CAD, particularly if they have a sibling younger than 60 years old who has premature CAD. Studies have shown that people who engage in regular, moderate intensity exercise can eliminate metabolic syndrome risk factors that can lead to CAD; however, many high-risk Black Americans do not take part in regular exercise. The purpose of this study is to compare a community-based, coach-led exercise program to an individual, self-led home-based exercise program to examine which program is more effective at reducing the metabolic syndrome risk factors that can lead to CAD in Black Americans.

This study will enroll Black Americans with metabolic syndrome who have a sibling with premature CAD. Participants will be randomly assigned (by individual) to either a community-based exercise program (C-FIT) or a self-help home-based exercise program (HOME). Participants in the C-FIT group will do 1 hour of exercise two to three times each week in a community setting and will be supervised by a personal coach or trainer for 1 year. Participants in the SELF group will undergo a fitness evaluation and will be instructed on how to exercise on their own. They also will be expected to do 1 hour of exercise two to three times each week for 1 year. Study visits will occur at baseline, Month 6, and Years 1 and 2. At all study visits, participants will undergo the following: a medical history review; physical examination; blood pressure measurements; blood collection; body measurements, including height, weight, and waist circumference; a treadmill stress test; a strength test; a dual-energy x-ray absorptiometry (DEXA) scan to measure body fat; an echocardiogram to examine the heart; a flow-mediated vasodilatation test for brachial reactivity to measure vascular function; and questionnaires on diet, exercise habits, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the Johns Hopkins Sibling and Family Heart Studies
* Has metabolic syndrome components
* Self-identifies as Black American

Exclusion Criteria:

* Any clinical CAD
* Diabetes
* Major co-morbidity that precludes exercise (e.g., stroke, AIDS, cancer, neurological disorder, serious emphysema or exercise asthma, disabling arthritis)
* Resting systolic blood pressure greater than or equal to 160 mm Hg, resting diastolic blood pressure greater than or equal to 100 mm Hg, or exercise peak blood pressure greater than or equal to 250/115 mm Hg
* Known ejection fraction less than 40%
* Already participating in regular exercise, defined as 90 minutes per week of activities of greater than 5 metabolic equivalents (METS)
* Cardiac arrhythmias, including supraventricular tachycardia in the 5 years before study entry, any ventricular tachycardia, or greater than 4-beat runs of nonsustained premature ventricular contractions on baseline screening exercise testing
* Body mass index (BMI) greater than 45 kg/m2
* Alcohol or substance abuse in the 12 months before study entry
* A known abnormal exercise electrocardiogram and an abnormal thallium scan (double abnormal), a moderate to severe defect on thallium scan, or a coronary calcium score greater than 500 on a prior screening
* An abnormal exercise screening test supervised by a physician as part of this study
* Pregnant
* Current smokers if they have stated evidence of shortness of breath with normal exercises or a diagnosis of chronic obstructive pulmonary disease by their physician, as verified by medical records

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in maximal oxygen consumption (VO2 max) | Measured at baseline, Month 6, and Years 1 and 2
Reduction in components of the metabolic syndrome | Measured at baseline and Years 1 and 2

SECONDARY OUTCOMES:
habitual physical activity score using a standardized questionnaire | 6 months, 1 year, 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Institute for Clinical Translational Research, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kral BG, Becker LC, Vaidya D, Yanek LR, Becker DM. Silent myocardial ischaemia and long-term coronary artery disease outcomes in apparently healthy people from families with early-onset ischaemic heart disease. Eur Heart J. 2011 Nov;32(22):2766-72. doi: 10.1093/eurheartj/ehr261. Epub 2011 Jul 23. PMID 21785111
- [Result] Brown RV, Kral BG, Yanek LR, Vaidya D, Nyquist PA, Levine DM, Moy TF, Becker LC, Becker DM. Ethnic-specific determinants of exercise capacity in a healthy high-risk population. Med Sci Sports Exerc. 2012 Jun;44(6):1150-6. doi: 10.1249/MSS.0b013e3182456990. PMID 22215178